CLINICAL TRIAL: NCT00700115
Title: A Pilot Study to Assess the Safety, Efficacy, and PK Profile of a Switch in Antiretroviral Therapy to a RTI Sparing Combination of LPV/r and RAL in Virologically Suppressed HIV-infected Patients
Brief Title: Kaletra-isentress Treatment Evaluation
Acronym: KITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Abbott (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ighovwerha Ofotokun, Associate Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006876; KITE-6876 (Other: Other)
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-11

CONDITIONS: HIV Infections
Keywords: HAART; lopinavir/ritonavir; raltegravir; HIV/AIDS patients on HAART; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Raltegravir Potassium; Lopinavir; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kaletra + Isentress (Experimental): Kaletra + Isentress
  Interventions: Drug: Kaletra + Isentress
- Standard HAART (Active Comparator): Pre-study Antiretroviral regimen
  Interventions: Drug: Pre-study antiretroviral regimen

INTERVENTIONS:
Drug: Kaletra + Isentress — Kaletra 400/100 mg + Isentress 400 mg BID
  Other Names: Raltegravir; Lopinavir/ritonavir
  Arms: Kaletra + Isentress
Drug: Pre-study antiretroviral regimen — Standard doses of pre-study antiretroviral regimen
  Other Names: HAART
  Arms: Standard HAART

SUMMARY:
This study will examine the effectiveness and safety of raltegravir (isentress) when used together with lopinavir/ritonavir (kaletra) for the treatment of HIV-infection. Isentress is a recently, Food and Drug Administration (FDA) approved, HIV medication that has strong effects against the HIV virus. Isentress has been shown in other studies to be safe and well tolerated by HIV patients. Combining this drug with kaletra might enable us to construct a HIV regimen that does not include the more toxic drugs of the nucleoside reverse transcriptase inhibitor class.

Eligible volunteers will undergo the following as part of the study procedure:

1. Sign the study consent form and the HIPAA Authorization Form.
2. Two-third of subjects, the intervention group (selected by random chance) will have their HIV drug treatment changed to kaletra + isentress.
3. The other one-third will continue their usual HIV medications (this will be the control group).
4. Make 9 study related visits to the Ponce clinic during the 48 weeks study period. During these visits, medical information will be collected, and blood tests will be performed.
5. Perform Dexa-scan on two separate occasions at Emory University Hospital Radiology.

Information collected will be used to assess the effectiveness of this treatment in keeping the HIV virus suppressed, how well these two drugs together is tolerated by HIV-infected patients, and the blood levels of these two drugs when given together.

DETAILED DESCRIPTION:
RATIONALE: Virologic failure and adverse effects associated with current highly active antiretroviral therapy (HAART) warrant continuing search for novel combination therapeutic options. Raltegravir's (RAL) was recently shown to be a potent antiretroviral (ARV) agent with a favorable safety profile. If future reports continue to show positive data on this first-in-class integrase inhibitor, there may be a paradigm shift in the currently recommended first line HAART to regimens that will include integrase inhibitors.

Combining RAL with a drug that has a high genetic barrier to resistance, such as lopinavir/ritonavir (LPV/r) may offer a number of advantages. Both agents are potent and should produce durable virologic suppression. Because their combination is reverse transcriptase inhibitor (RTI) class sparing, its tolerability might be superior. In addition, RAL is not metabolized by the cytochrome P-450 enzymes, therefore, a compatible pharmacokinetic profile is expected with this combination. Pairing LPV/r with RAL in early ARV regimens as is proposed in this application may provide a HAART regimen that is highly efficacious and durable, with less resistance and adverse drug events.

DESIGN: This is single center, open label, randomized, controlled, study designed to assess the tolerability, pharmacokinetic compatibility, and the durability of virologic suppression of the RTI sparing combination therapy of LPV/r + RAL. HIV-infected subjects who are virologically suppressed (HIV-RNA PCR < 50 copies/ml) on current HAART regimen will be randomized in a 2:1 fashion to be switched to a regimen consisting of LPV/r + RAL, intervention arm A (n=40), or to be continued on their pre-study HAART regimen, control arm B (n=20). The primary endpoint will be proportion of subjects with sustained virologic suppression (HIV-1 RNA PCR < 50 copies/ml) through week 48. The immunoreconstitution, toxicity profile, and pharmacokinetic profile of the RAL and LPV/r in this novel combination therapy will be evaluated.

DURATION: 48 weeks after the enrollment of the last participant. Enrollment is expected to take about 10 months.

SAMPLE SIZE: 60 subjects.

POPULATION: HIV-infected individuals (male and female), Age > 18 years, who are virologically suppressed (HIV-RNA PCR < 50 copies/ml) on their current HAART regimen for > 6 months.

REGIMEN: For Arm A= LPV/r 400/100 mg (2 tablets) twice daily + RAL 400 mg (1 tablet) twice daily taken by mouth. For Arm B=Pre-study HAART regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected individuals receiving HAART regimen (if on PI-based regimen, must be 1st PI-containing HAART).
* They must have been on and tolerating current HAART regimen for > 6-months.
* Plasma HIV-1 viral load < 50 copies/ml at study entry.
* Men and women age > 18 years (sex is defined as sex at birth).
* Laboratory values obtained within 30 days prior to study entry:

  * Hemoglobin > 9.4 g/dl
  * Creatinine < 2 mg/dl
  * AST (SGOT) < 2 x ULN
  * ALT (SGPT) < 2 x ULN
* Ability and willingness of subject or legal guardian/representative to give written informed consent.
* No CD4 T-cell counts requirement

Exclusion Criteria:

* Subjects with a history of previous intolerance to or virological failure to LPV/r
* Concomitant drugs (including alternative therapies) that may affect PI or RAL plasma concentrations (inducers or inhibitors of the CYP 3A4 or UDP-glucuronosyltransferase iso-enzymes).
* A known history of noncompliance with medications or a known history of noncompliance with scheduled physician and clinic visits.
* Investigational ARV drug.
* Pregnancy/Breast feeding.
* HBV-coinfected patients receiving nucleoside analogue for both HIV and HBV suppression.
* Active drug or alcohol use or dependence which, in the Investigator's opinion, may interfere with adherence to study requirements or endanger subject's health while on the study.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igho Ofotokun, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Infectious Diseases Program (Ponce Clinic), Atlanta, Georgia, United States

REFERENCES:
- [Result] Ofotokun I, Sheth AN, Sanford SE, Easley KA, Shenvi N, White K, Eaton ME, Del Rio C, Lennox JL. A switch in therapy to a reverse transcriptase inhibitor sparing combination of lopinavir/ritonavir and raltegravir in virologically suppressed HIV-infected patients: a pilot randomized trial to assess efficacy and safety profile: the KITE study. AIDS Res Hum Retroviruses. 2012 Oct;28(10):1196-206. doi: 10.1089/AID.2011.0336. Epub 2012 Apr 20. PMID 22364141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from an urban outpatient HIV clinic (the Grady Infectious Diseases Program Out-patient Clinic, Atlanta, Georgia) between June 2008 and January 2011.
Pre-assignment Details: Subjects were excluded if they were on medications that could interact with Protease inhibitors, had an active opportunistic infection, had renal and/or hepatic impairment, or were pregnant. Hepatitis B virus (HBV) co-infected patients receiving a nucleotide analogue for both HIV and HBV suppression were also excluded from enrollment.
Groups:
- Kaletra + Isentress: Switched to Kaletra + Isentress
- Standard HAART: Pre-study standard HAART regimen
Period: Overall Study
Arm/Group | Kaletra + Isentress | Standard HAART
Started | 40 | 20
Completed | 39 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kaletra + Isentress | Standard HAART | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 20 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9) | 48 (12) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 26 | 12 | 38
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60

OUTCOME MEASURES:

1. Secondary Outcome: To Compare Plasma Triglyceride Levels at 48 Weeks Between LPV/r + RAL and Standard HAART Treated Subjects
Time Frame: 48 weeks
Population: intention to treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Kaletra + Isentress | Standard HAART
Number analyzed (Participants) | 35 | 19
mg/dL | 238.1 (19.9) | 133.3 (27.1)

2. Primary Outcome: Plasma Viral Loads (HIV-1 RNA PCR)
Description: Percentage subjects with undetectable Plasma viral loads
Time Frame: baseline to week 48
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Kaletra + Isentress | Standard HAART
Number analyzed (Participants) | 40 | 20
percentage of subjects | 92.7 [83 to 100] | 88 [75 to 100]

ADVERSE EVENTS:
Arm/Group | Kaletra + Isentress | Standard HAART
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/19
Other Adverse Events (participants affected / at risk) | 0/39 | 0/19

LIMITATIONS AND CAVEATS:
The findings of the KITE study should be interpreted in the context of a pilot study with a small sample size. Furthermore, adverse effects were self-reported, and the lack of blinding may have introduced biases in the collection of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No